CLINICAL TRIAL: NCT01614574
Title: A Multicenter, Open-Label Study of Velaglucerase Alfa Enzyme Replacement Therapy in Japanese Patients With Gaucher Disease
Brief Title: Study of Velaglucerase Alfa Enzyme Replacement Therapy in Japanese Patients With Gaucher Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGT-GCB-087
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease | interventions — Glucosylceramidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Investigational (Experimental): velaglucerase alfa
  Interventions: Biological: velaglucerase alfa

INTERVENTIONS:
Biological: velaglucerase alfa — 60 U/kg every other week intravenous infusion
  Other Names: VPRIV; Gene activated human glucocerebrosidase

SUMMARY:
Gaucher disease is an inherited deficiency of the lysosomal enzyme glucocerebrosidase (GCB) that leads to progressive accumulation of glucocerebroside within macrophages and subsequent tissue and organ damage; typically of the liver, spleen, bone marrow, and brain. The disease has been classified into 3 clinical subtypes based on the presence or absence of neurological symptoms and severity of neurological disease. Type 1 Gaucher disease affects an estimated 30,000 persons worldwide and is the most common. Type 1 Gaucher disease does not involve the central nervous system. Patients with type 2 Gaucher disease present with acute neurological deterioration, which leads to early death. Those with type 3 disease typically display a more sub-acute neurological course, with later onset and slower progression.

The primary objective of this study is to evaluate the safety of every other week dosing of velaglucerase alfa in Japanese patients with Gaucher disease.

Velaglucerase alfa has been developed and approved as an enzyme replacement therapy for Type 1 Gaucher disease.

DETAILED DESCRIPTION:
Gaucher disease is an inherited deficiency of the lysosomal enzyme glucocerebrosidase (GCB) that leads to progressive accumulation of glucocerebroside within macrophages and subsequent tissue and organ damage; typically of the liver, spleen, bone marrow, and brain.

Gaucher disease has been designated in the list of Specified Rare and Intractable Diseases by Specified Disease Treatment Research Program of Ministry of Health, Labor and Welfare (MHLW) as one of "lysosomal storage diseases" since 2001. Gaucher disease is also designated in the Medical Aid Program for Specified Categories of Chronic Pediatric Diseases.

The prevalence of mutations and the phenotype of patients with Gaucher disease in Japan differs from that in non-Japanese populations. Some patients with type 1 Gaucher disease in Japan have more severe and progressive disease compared to non-Japanese patients and the disease is characterized by an earlier onset of symptoms.

Velaglucerase alfa, a highly-purified form of the naturally occurring enzyme glucocerebrosidase, has been developed as an enzyme replacement therapy for Gaucher disease for the symptoms (anemia, thrombocytopenia, hepatomegaly, splenomegaly, and bone manifestation).

The primary objective of this study is to evaluate the safety of every other week dosing of velaglucerase alfa in Japanese patients (naive or previously treated with imiglucerase) 2 years of age and older with Gaucher disease.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a documented diagnosis of Gaucher disease
* The patient is at least 2 years of age
* Female patients of child bearing potential must agree to use a medically acceptable method of contraception at all times during the study
* The patient, the patient's parent(s) or legal guardian(s) has provided written informed consent that has been approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC)
* The patient must be sufficiently cooperative to participate in this clinical study as judged by the Investigator

Patients who are switched from imiglucerase ERT must meet the following additional criteria:

* Received treatment with imiglucerase for a minimum of 12 consecutive months
* Meet predefined limits for hemoglobin concentration and platelet counts

Patients naïve to treatment for Gaucher disease must meet the following additional criteria:

* Not received treatment for Gaucher disease (investigational or approved products) within 12 months prior to study entry
* Have Gaucher disease related anemia and at least one of the following: moderate splenomegaly or, Gaucher disease-related thrombocytopenia or Gaucher disease-related enlarged liver

Exclusion Criteria:

* Treatment with any investigational drug or device within the 30 days prior to study entry (time of informed consent); such use during the study is not permitted
* Positive for hepatitis B or hepatitis C.
* Non-Gaucher disease related anemia
* The patient, patient's parent(s), or patient's legal guardian(s) is/are unable to understand the nature, scope, and possible consequences of the study
* Significant comorbidity, as determined by the Investigator that might affect study data or confound the study results
* The patient is unable to comply with the protocol or is unlikely to complete the study, as determined by the Investigator
* The patient has experienced a severe (grade 3 or higher) infusion-related hypersensitivity reaction (anaphylactic or anaphylactoid reaction) to any ERT (approved or investigational)
* Currently receiving red blood cell growth factor, (eg, erythropoietin) or chronic systemic corticosteroids in the last 6 months
* Patient has had a splenectomy or the patient has an active, clinically significant spleen infarction within 12 months of screening
* Patient has worsening bone necrosis within 12 months of screening
* The patient is pregnant or lactating.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-03-02 (Actual); Primary Completion 2013-05-25 (Actual); Study Completion 2013-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- Japan (3):
  - Hamamatsu University School of Medicine, Hamamatsu, Shizuoka
  - The Jikei University School of Medicine, Minatoku, Toyko
  - Osaka City University Hospital, Osaka

RESULTS

PARTICIPANT FLOW:
Groups:
- VPRIV® (15-60 U/kg): Administered as an intravenous (IV) infusion over a 60 minute period.
Period: Overall Study
Arm/Group | VPRIV® (15-60 U/kg)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VPRIV® (15-60 U/kg)
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20 (10.62)
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Count of Participants; unit: Participants]
  JAPAN | 6
Hemoglobin Concentration [Mean (Standard Deviation); unit: (g/dL)] | 13.77 (0.954)
Platelet Count [Mean (Standard Deviation); unit: (x 10^9 platelets/L)] | 182.9 (32.05)
Normalized liver volume [Mean (Standard Deviation); unit: (% of Body Weight)] | 1.92 (0.342)
Normalized spleen volume [Mean (Standard Deviation); unit: (% of Body Weight)] | 0.39 (0.067)
Plasma chitotriosidase [Mean (Standard Deviation); unit: (nmol/mL/h)] | 1243.7 (344.46)
CCL18 levels [Mean (Standard Deviation); unit: (ng/mL)] | 134.8 (132.26)

OUTCOME MEASURES:

1. Primary Outcome: Number of Severe Adverse Events (SAE)
Time Frame: Baseline to week 51
Measure: Number; unit: events
Arm/Group | VPRIV® (15-60 U/kg)
Number analyzed (Participants) | 6
events | 1

2. Primary Outcome: Number of Treatment Emergent Adverse Events (TEAE)
Time Frame: Baseline to week 51
Measure: Number; unit: events
Arm/Group | VPRIV® (15-60 U/kg)
Number analyzed (Participants) | 6
events | 31

3. Primary Outcome: Development of Anti-velaglucerase Alfa Antibody
Time Frame: Baseline to week51
Measure: Number; unit: participants
Arm/Group | VPRIV® (15-60 U/kg)
Number analyzed (Participants) | 6
participants
  Positive (Baseline) | 0
  Negative (Baseline) | 6
  Positive (Week 51) | 0
  Negative (Week 51) | 6

4. Primary Outcome: Number of Infusion- Related Adverse Events
Time Frame: Baseline to week 51
Measure: Number; unit: events
Arm/Group | VPRIV® (15-60 U/kg)
Number analyzed (Participants) | 6
events | 2

5. Primary Outcome: Number of Patients With Concomitant Medication
Time Frame: Baseline to week 51
Measure: Number; unit: participants
Arm/Group | VPRIV® (15-60 U/kg)
Number analyzed (Participants) | 6
participants | 6

6. Secondary Outcome: Change From Baseline in Hemoglobin Concentration
Time Frame: Baseline to week 51
Measure: Mean (Standard Deviation); unit: (g/dL)
Arm/Group | VPRIV® (15-60 U/kg)
Number analyzed (Participants) | 6
(g/dL) | 0.05 (0.729)

7. Secondary Outcome: Change From Baseline in Platelet Count
Time Frame: Baseline to week 51
Measure: Mean (Standard Deviation); unit: (x 10^9 platelets/L)
Arm/Group | VPRIV® (15-60 U/kg)
Number analyzed (Participants) | 6
(x 10^9 platelets/L) | 13.8 (35.75)

8. Secondary Outcome: Change From Baseline in Liver Volume, Normalized to Body Weight
Time Frame: Baseline to week 51
Measure: Mean (Standard Deviation); unit: (% of Body Weight)
Arm/Group | VPRIV® (15-60 U/kg)
Number analyzed (Participants) | 6
(% of Body Weight) | 0.05 (0.148)

9. Secondary Outcome: Change From Baseline in Spleen Volume, Normalized to Body Weight
Time Frame: Baseline to week 51
Measure: Mean (Standard Deviation); unit: (% of Body Weight)
Arm/Group | VPRIV® (15-60 U/kg)
Number analyzed (Participants) | 6
(% of Body Weight) | 0.39 (0.067)

10. Secondary Outcome: Change From Baseline in Plasma Chitotriosidase Levels
Time Frame: Baseline to week 51
Measure: Mean (Standard Deviation); unit: (nmol/mL/h)
Arm/Group | VPRIV® (15-60 U/kg)
Number analyzed (Participants) | 6
(nmol/mL/h) | -47.3 (64.44)

11. Secondary Outcome: Change From Baseline in CCL18 Levels
Time Frame: Baseline to week 51
Measure: Mean (Standard Deviation); unit: (ng/mL)
Arm/Group | VPRIV® (15-60 U/kg)
Number analyzed (Participants) | 6
(ng/mL) | 5.2 (10.59)

ADVERSE EVENTS:
Arm/Group | VPRIV® (15-60 U/kg)
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VPRIV® (15-60 U/kg) (N=6)
RETINAL DETACHMENT (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VPRIV® (15-60 U/kg) (N=6)
RETINOPATHY PROLIFERATIVE (Eye disorders) | 1 (1)
VISUAL ACUITY REDUCED (Eye disorders) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1)
CHEILITIS (Gastrointestinal disorders) | 1 (1)
ENTERITIS (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 1 (1)
SUBMANDIBULAR MASS (General disorders) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (2)
HAND-FOOT-AND-MOUTH DISEASE (Infections and infestations) | 1 (1)
HORDEOLUM (Infections and infestations) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 6 (9)
OTITIS MEDIA (Infections and infestations) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 3 (3)
JOINT SPRAIN (Injury, poisoning and procedural complications) | 1 (1)
LIMB INJURY (Injury, poisoning and procedural complications) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
HEADACHE (Nervous system disorders) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1)
MYOCLONUS (Nervous system disorders) | 1 (1)
ADJUSTMENT DISORDER (Psychiatric disorders) | 1 (1)
MENSTRUATION IRREGULAR (Reproductive system and breast disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (2)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1)
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ACNE (Skin and subcutaneous tissue disorders) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
All 6 enrolled patients received previous long-term treatment with the enzyme replacement therapy (ERT), imiglucerase. Key therapeutic parameters were expected to indicate stability after switching from imiglucerase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Shire's agreements with investigators vary. All agreements provide Shire the right to embargo communications regarding trial results prior to public release for a period ≤180 days from the time submitted to Shire for review. Shire does not prohibit publication, but can require the removal of confidential information (excluding trial results) and can request postponement of a single-center publication until after disclosure of the trial's multi-center publication